CLINICAL TRIAL: NCT02541864
Title: Comparison of Hybrid and Bismuth Containing Quadruple Therapies for Helicobacter Pylori Eradication: a Randomized Controlled Trial
Brief Title: Comparison of Hybrid and Bismuth Quadruple Therapies for Helicobacter Pylori Eradication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Feng-Woei Tsay, ASSISTANT PROFESSOR, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS12-CT11-08
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2015-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Hybrid therapy; Bismuth containing quadruple therapy; Eradication
MeSH Terms: interventions — Pantoprazole; bismuth tripotassium dicitrate; Tetracycline; Metronidazole; Hybrid Renal Replacement Therapy; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bismuth quadruple therapy (Experimental): pantoprazole 40 mg bid for 14 days, bismuth subcitrate 120 mg qid for 14 days, tetracycline 500 mg qid for 14 days, metronidazole 250 mg qid for 14 days
  Interventions: Drug: Bismuth quadruple therapy
- Hybrid therapy (Active Comparator): (pantoprazole 40 mg bid for 7 days, amoxicillin 1 g bid for 7 days) followed by (pantoprazole 40 mg bid for 7 days, amoxicillin 1 g bid for 7 days, clarithromycin 500 mg bid for 7 days, and metronidazole 500 mg bid for 7 days)
  Interventions: Drug: Hybrid therapy

INTERVENTIONS:
Drug: Bismuth quadruple therapy — pantoprazole 40 mg bid for 14 days, bismuth subcitrate 120 mg qid for 14 days, tetracycline 500 mg qid for 14 days, metronidazole 250 mg qid for 14 days
  Other Names: pantoprazole; bismuth subcitrate; tetracycline; metronidazole
  Arms: Bismuth quadruple therapy
Drug: Hybrid therapy — (pantoprazole 40 mg bid for 7 days, amoxicillin 1 g bid for 7 days) followed by (pantoprazole 40 mg bid for 7 days, amoxicillin 1 g bid for 7 days, clarithromycin 500 mg bid for 7 days, and metronidazole 500 mg bid for 7 days)
  Other Names: pantoprazole; amoxicillin; clarithromycin; metronidazole
  Arms: Hybrid therapy

SUMMARY:
According the Maastricht IV consensus report publish in the Gut 2012, bismuth containing quadruple therapy was suggested to be the first choice for eradication therapy of Helicobacter pylori in the area with high clarithromycin resistance. Whether hybrid therapy or 14-day bismuth containing quadruple therapy can replace standard triple therapy as the recommended first-line treatment is unknown. The investigators compared the efficacy of 14-day hybrid therapy and 14-day bismuth containing quadruple therapy in first-line treatment.

DETAILED DESCRIPTION:
For this randomly assigned to receive either a 14-day hybrid therapy (a dual therapy with pantoprazole 40 mg bid, amoxicillin 1 g bid for 7 days, followed by a quadruple therapy with pantoprazole 40 mg bid, amoxicillin 1 g bid, clarithromycin 500 mg bid, and metronidazole 500 mg bid for a further 7 days) or a 14-day bismuth containing quadruple therapies (pantoprazole 40 mg bid , bismuth subcitrate 120 mg qid., tetracycline 500 mg qid, and metronidazole 250 mg qid for 14 days).at a 1:1 ratio. Our primary outcomes was the eradication rate by intention-to-treat and per- protocol analyses

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H pylori-infected outpatients, at least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H pylori-eradication therapy
* ingestion of antibiotics or bismuth within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.

REFERENCES:
- [Background] Vakil N, Megraud F. Eradication therapy for Helicobacter pylori. Gastroenterology. 2007 Sep;133(3):985-1001. doi: 10.1053/j.gastro.2007.07.008. PMID 17854602
- [Background] Hunt RH, Lam SK. Helicobacter pylori: from art to a science. J Gastroenterol Hepatol. 1998 Jan;13(1):21-8. doi: 10.1111/j.1440-1746.1998.tb00540.x. PMID 9737567
- [Background] Graham DY, Lew GM, Klein PD, Evans DG, Evans DJ Jr, Saeed ZA, Malaty HM. Effect of treatment of Helicobacter pylori infection on the long-term recurrence of gastric or duodenal ulcer. A randomized, controlled study. Ann Intern Med. 1992 May 1;116(9):705-8. doi: 10.7326/0003-4819-116-9-705. PMID 1558340
- [Background] Sung JJ, Chung SC, Ling TK, Yung MY, Leung VK, Ng EK, Li MK, Cheng AF, Li AK. Antibacterial treatment of gastric ulcers associated with Helicobacter pylori. N Engl J Med. 1995 Jan 19;332(3):139-42. doi: 10.1056/NEJM199501193320302. PMID 7800005
- [Background] Hsu PI, Lai KH, Tseng HH, Lo GH, Lo CC, Lin CK, Cheng JS, Chan HH, Ku MK, Peng NJ, Chien EJ, Chen W, Hsu PN. Eradication of Helicobacter pylori prevents ulcer development in patients with ulcer-like functional dyspepsia. Aliment Pharmacol Ther. 2001 Feb;15(2):195-201. doi: 10.1046/j.1365-2036.2001.00903.x. PMID 11148437
- [Background] Satoh K. Does eradication of Helicobacter pylori reverse atrophic gastritis or intestinal metaplasia? Data from Japan. Gastroenterol Clin North Am. 2000 Dec;29(4):829-35. doi: 10.1016/s0889-8553(05)70150-3. PMID 11190067
- [Background] Isaacson PG. Recent developments in our understanding of gastric lymphomas. Am J Surg Pathol. 1996;20 Suppl 1:S1-7. doi: 10.1097/00000478-199600001-00002. PMID 8694145
- [Background] Wong BC, Lam SK, Wong WM, Chen JS, Zheng TT, Feng RE, Lai KC, Hu WH, Yuen ST, Leung SY, Fong DY, Ho J, Ching CK, Chen JS; China Gastric Cancer Study Group. Helicobacter pylori eradication to prevent gastric cancer in a high-risk region of China: a randomized controlled trial. JAMA. 2004 Jan 14;291(2):187-94. doi: 10.1001/jama.291.2.187. PMID 14722144
- [Background] Malfertheiner P, Megraud F, O'Morain C, Bazzoli F, El-Omar E, Graham D, Hunt R, Rokkas T, Vakil N, Kuipers EJ. Current concepts in the management of Helicobacter pylori infection: the Maastricht III Consensus Report. Gut. 2007 Jun;56(6):772-81. doi: 10.1136/gut.2006.101634. Epub 2006 Dec 14. PMID 17170018
- [Background] Hsu PI, Lai KH, Lin CK, Chen WC, Yu HC, Cheng JS, Tsay FW, Wu CJ, Lo CC, Tseng HH, Yamaoka Y, Chen JL, Lo GH. A prospective randomized trial of esomeprazole- versus pantoprazole-based triple therapy for Helicobacter pylori eradication. Am J Gastroenterol. 2005 Nov;100(11):2387-92. doi: 10.1111/j.1572-0241.2005.00264.x. PMID 16279889
- [Background] Wu IC, Wu DC, Hsu PI, Lu CY, Yu FJ, Wang TE, Chang WH, Chen JJ, Kuo FC, Wu JY, Wang WM, Bair MJ. Rabeprazole- versus esomeprazole-based eradication regimens for H. pylori infection. Helicobacter. 2007 Dec;12(6):633-7. doi: 10.1111/j.1523-5378.2007.00553.x. PMID 18001406
- [Background] Fock KM, Katelaris P, Sugano K, Ang TL, Hunt R, Talley NJ, Lam SK, Xiao SD, Tan HJ, Wu CY, Jung HC, Hoang BH, Kachintorn U, Goh KL, Chiba T, Rani AA; Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol. 2009 Oct;24(10):1587-600. doi: 10.1111/j.1440-1746.2009.05982.x. PMID 19788600
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Graham DY, Lu H, Yamaoka Y. Therapy for Helicobacter pylori infection can be improved: sequential therapy and beyond. Drugs. 2008;68(6):725-36. doi: 10.2165/00003495-200868060-00001. PMID 18416582
- [Background] Gumurdulu Y, Serin E, Ozer B, Kayaselcuk F, Ozsahin K, Cosar AM, Gursoy M, Gur G, Yilmaz U, Boyacioglu S. Low eradication rate of Helicobacter pylori with triple 7-14 days and quadriple therapy in Turkey. World J Gastroenterol. 2004 Mar 1;10(5):668-71. doi: 10.3748/wjg.v10.i5.668. PMID 14991935
- [Background] Bigard MA, Delchier JC, Riachi G, Thibault P, Barthelemy P. One-week triple therapy using omeprazole, amoxycillin and clarithromycin for the eradication of Helicobacter pylori in patients with non-ulcer dyspepsia: influence of dosage of omeprazole and clarithromycin. Aliment Pharmacol Ther. 1998 Apr;12(4):383-8. doi: 10.1046/j.1365-2036.1998.00315.x. PMID 9690730
- [Background] Graham DY, Shiotani A. New concepts of resistance in the treatment of Helicobacter pylori infections. Nat Clin Pract Gastroenterol Hepatol. 2008 Jun;5(6):321-31. doi: 10.1038/ncpgasthep1138. Epub 2008 Apr 29. PMID 18446147
- [Background] Chuah SK, Tsay FW, Hsu PI, Wu DC. A new look at anti-Helicobacter pylori therapy. World J Gastroenterol. 2011 Sep 21;17(35):3971-5. doi: 10.3748/wjg.v17.i35.3971. PMID 22046084
- [Background] Zullo A, Vaira D, Vakil N, Hassan C, Gatta L, Ricci C, De Francesco V, Menegatti M, Tampieri A, Perna F, Rinaldi V, Perri F, Papadia C, Fornari F, Pilati S, Mete LS, Merla A, Poti R, Marinone G, Savioli A, Campo SM, Faleo D, Ierardi E, Miglioli M, Morini S. High eradication rates of Helicobacter pylori with a new sequential treatment. Aliment Pharmacol Ther. 2003 Mar 1;17(5):719-26. doi: 10.1046/j.1365-2036.2003.01461.x. PMID 12641522
- [Background] Vaira D, Zullo A, Vakil N, Gatta L, Ricci C, Perna F, Hassan C, Bernabucci V, Tampieri A, Morini S. Sequential therapy versus standard triple-drug therapy for Helicobacter pylori eradication: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):556-63. doi: 10.7326/0003-4819-146-8-200704170-00006. PMID 17438314
- [Background] Gatta L, Vakil N, Leandro G, Di Mario F, Vaira D. Sequential therapy or triple therapy for Helicobacter pylori infection: systematic review and meta-analysis of randomized controlled trials in adults and children. Am J Gastroenterol. 2009 Dec;104(12):3069-79; quiz 1080. doi: 10.1038/ajg.2009.555. Epub 2009 Oct 20. PMID 19844205
- [Background] Sanchez-Delgado J, Calvet X, Bujanda L, Gisbert JP, Tito L, Castro M. Ten-day sequential treatment for Helicobacter pylori eradication in clinical practice. Am J Gastroenterol. 2008 Sep;103(9):2220-3. doi: 10.1111/j.1572-0241.2008.01924.x. Epub 2008 Jun 28. PMID 18564109
- [Background] Tsay FW, Tseng HH, Hsu PI, Wang KM, Lee CC, Chang SN, Wang HM, Yu HC, Chen WC, Peng NJ, Lai KH, Wu DC. Sequential therapy achieves a higher eradication rate than standard triple therapy in Taiwan. J Gastroenterol Hepatol. 2012 Mar;27(3):498-503. doi: 10.1111/j.1440-1746.2011.06885.x. PMID 21871025
- [Background] Choi WH, Park DI, Oh SJ, Baek YH, Hong CH, Hong EJ, Song MJ, Park SK, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI. [Effectiveness of 10 day-sequential therapy for Helicobacter pylori eradication in Korea]. Korean J Gastroenterol. 2008 May;51(5):280-4. Korean. PMID 18516011
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Background] Greenberg ER, Anderson GL, Morgan DR, Torres J, Chey WD, Bravo LE, Dominguez RL, Ferreccio C, Herrero R, Lazcano-Ponce EC, Meza-Montenegro MM, Pena R, Pena EM, Salazar-Martinez E, Correa P, Martinez ME, Valdivieso M, Goodman GE, Crowley JJ, Baker LH. 14-day triple, 5-day concomitant, and 10-day sequential therapies for Helicobacter pylori infection in seven Latin American sites: a randomised trial. Lancet. 2011 Aug 6;378(9790):507-14. doi: 10.1016/S0140-6736(11)60825-8. Epub 2011 Jul 21. PMID 21777974
- [Background] Hsu PI, Wu DC, Wu JY, Graham DY. Modified sequential Helicobacter pylori therapy: proton pump inhibitor and amoxicillin for 14 days with clarithromycin and metronidazole added as a quadruple (hybrid) therapy for the final 7 days. Helicobacter. 2011 Apr;16(2):139-45. doi: 10.1111/j.1523-5378.2011.00828.x. PMID 21435092
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Hsu PI, Lai KH, Wu CJ, Tseng HH, Tsay FW, Peng NJ, Chen TA, Chuah SK, Lin WS, Lo GH. High-dose versus low-dose esomeprazole-based triple therapy for Helicobacter pylori infection. Eur J Clin Invest. 2007 Sep;37(9):724-30. doi: 10.1111/j.1365-2362.2007.01852.x. PMID 17696962
- [Background] Hsu PI, Lai KH, Tseng HH, Liu YC, Yen MY, Lin CK, Lo GH, Huang RL, Huang JS, Cheng JS, Huang WK, Ger LP, Chen W, Hsu PN. Correlation of serum immunoglobulin G Helicobacter pylori antibody titers with histologic and endoscopic findings in patients with dyspepsia. J Clin Gastroenterol. 1997 Dec;25(4):587-91. doi: 10.1097/00004836-199712000-00007. PMID 9451668
- [Background] Dixon MF, Genta RM, Yardley JH, Correa P. Classification and grading of gastritis. The updated Sydney System. International Workshop on the Histopathology of Gastritis, Houston 1994. Am J Surg Pathol. 1996 Oct;20(10):1161-81. doi: 10.1097/00000478-199610000-00001. PMID 8827022
- [Background] Hsu PI, Wu DC, Wu JY, Graham DY. Is there a benefit to extending the duration of Helicobacter pylori sequential therapy to 14 days? Helicobacter. 2011 Apr;16(2):146-52. doi: 10.1111/j.1523-5378.2011.00829.x. PMID 21435093
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Clinical significance of oral urease in diagnosis of Helicobacter pylori infection by [13C]urea breath test. Dig Dis Sci. 2001 Aug;46(8):1772-8. doi: 10.1023/a:1010626225949. PMID 11508681
- [Derived] Tsay FW, Wu DC, Yu HC, Kao SS, Lin KH, Cheng JS, Wang HM, Chen WC, Sun WC, Tsai KW, Hsu PI. A Randomized Controlled Trial Shows that both 14-Day Hybrid and Bismuth Quadruple Therapies Cure Most Patients with Helicobacter pylori Infection in Populations with Moderate Antibiotic Resistance. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e00140-17. doi: 10.1128/AAC.00140-17. Print 2017 Nov. PMID 28807915

RESULTS

PARTICIPANT FLOW:
Groups:
- Pantoprazole+Bismuth+Tetra+Metro: pantoprazole 40 mg bid , bismuth subcitrate 120 mg qid., tetracycline 500 mg qid, metronidazole 250 mg qid for 14 days
  pantoprazole+bismuth+tetra+metro: pantoprazole 40 mg bid , bismuth subcitrate 120 mg qid., tetracycline 500 mg qid, and metronidazole 250 mg qid for 14 days
- Hybrid Therapy: a dual therapy with pantoprazole 40 mg bid, amoxicillin 1 g bid for 7 days, followed by a quadruple therapy with pantoprazole 40 mg bid, amoxicillin 1 g bid, clarithromycin 500 mg bid, and metronidazole 500 mg bid for a further 7 days
  Hybrid therapy: a dual therapy with pantoprazole 40 mg bid, amoxicillin 1 g bid for 7 days, followed by a quadruple therapy with pantoprazole 40 mg bid, amoxicillin 1 g bid, clarithromycin 500 mg bid, and metronidazole 500 mg bid for a further 7 days
Period: Overall Study
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | Hybrid Therapy
Started | 164 | 166
Completed | 164 | 166
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | Hybrid Therapy | Total
Number analyzed (Participants) | 164 | 166 | 330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 134 | 136 | 270
  >=65 years | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.46 (12.28) | 54.48 (11.45) | 53.97 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 87 | 157
  Male | 94 | 79 | 173
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 164 | 166 | 330

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: Repeated endoscopy with rapid urease test, histological examination and culture or urea breath tests are conducted to assess H. pylori status.
Time Frame: at the 6th week after the end of anti- H. pylori therapy
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | Hybrid Therapy
Number analyzed (Participants) | 164 | 166
participants | 154 | 154

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | Hybrid Therapy
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/166
Other Adverse Events (participants affected / at risk) | 92/164 | 19/166
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole+Bismuth+Tetra+Metro (N=164) | Hybrid Therapy (N=166)
Nausea (Gastrointestinal disorders) | 75 (75) | 12 (12) — Patients had Nausea discomforts.
Dizziness (Gastrointestinal disorders) | 17 (17) | 7 (7) — Patients had dizziness discomforts.

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes